CLINICAL TRIAL: NCT04483466
Title: Methotrexate Treatment of Arthritis Caused by Chikungunya Virus (MARCH): A Phase III Randomized Controlled Clinical Trial of the Efficacy of Methotrexate Monotherapy in the Treatment of Chronic Arthritis After Chikungunya Infection
Brief Title: Methotrexate Treatment of Arthritis Caused by Chikungunya Virus (MARCH)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Aileen Y Chang, Associate Professor of Medicine, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Chang_MARCH_JUNE2020
Record Dates: First submitted 2020-06-23; First posted 2020-07-23 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Investigate the Effect(s) of Methotrexate Treatment on Arthritis Disease Severity
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Intervention Model Description: * In the treatment group, participants will receive methotrexate 15mg by mouth/week with optional for increase up to 20mg/week in non-responders and folic acid 1mg by mouth daily for six months in Phase I.
  * In the control group, participants will receive placebo methotrexate tablets by mouth/week with faux increase optional in non-responders and folic acid 1mg by mouth daily for six months in Phase I.
  * In Phase II, any patient may elect to stop taking the study drug or transition to open label active treatment group for the following six months if non-responder.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment with methotrexate (Experimental): 100 participants will be treated with methotrexate
  Interventions: Drug: Methotrexate
- Placebo methotrexate (Placebo Comparator): 50 will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — Methotrexate is vibrant yellow-orange colored powder with physical properties of near insolubility in water formulated into methotrexate tablets containing an amount of methotrexate sodium equivalent to 2.5 mg of methotrexate and are round, convex, and yellow. The chemical name is N-[4-[[(2,4-diamino-6pteridinyl)methyl]methyl amino]benzoyl]-L-glutamic acid. Methotrexate is an anti-metabolite that is a folate antagonist that inhibits lymphocyte proliferation and functions as an immunosuppressant in arthritis.
  Arms: Treatment with methotrexate
Drug: Placebo — Placebo
  Arms: Placebo methotrexate

SUMMARY:
MARCH is the first randomized, double-blind, placebo-controlled evaluation of the efficacy and pathologic mechanism determined by synovial biopsy of 6 months of methotrexate (n=100) versus placebo (n=50) therapy for chronic chikungunya (CHIKV) arthritis in Colombia with the option for open-label use of the medication for up to one year for all participants. Our central hypothesis is that methotrexate will significantly decrease chronic CHIKV arthritis disease severity compared to placebo via suppression of leukocyte accumulation in synovial tissue and decreased expression of inflammatory cytokines from synovial macrophages and fibroblast-like synoviocytes (FLS).

DETAILED DESCRIPTION:
* In the treatment group, participants will receive methotrexate 15mg by mouth/week with optional for increase up to 20mg/week in non-responders and folic acid 1mg by mouth daily for six months in Phase I.
* In the control group, participants will receive placebo methotrexate tablets by mouth/week with faux increase optional in non-responders and folic acid 1mg by mouth daily for six months in Phase I.
* In Phase II, patients may elect to stop taking the study drug or in those without clinical remission transition to open label active treatment group for the following six months.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged >18 years
4. Ability to take oral medication and be willing to adhere to the methotrexate regimen
5. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 3 months after the end of methotrexate administration.
6. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner.
7. Have a diagnosis of CHIKV by CHIKV IgM or IgG antibody.
8. The disease duration should be greater than 3 months (based on onset of symptoms).
9. Screen laboratory tests must meet the following criteria: Hemoglobin ≥ 9 g/dL, WBCs ≥ 3.5 x 109 cells/L, Neutrophils ≥ 1.5 x 109 cells/L, Platelets ≥ 100 x 109 cells/L, serum transaminase levels not exceeding 1.5 times the upper limit of normal, serum creatinine ≤ 1.6 mg/dL, and negative for hepatitis B surface antigen and hepatitis C antibodies.
10. Have a chest radiograph at screening that shows no clear evidence of malignancy or active infection.
11. Have active moderate arthritis defined as at least 4 tender joints and at least one joint with definite clinical synovitis (swelling). Joints that may be considered in the count include the temporomandibular joints (0-2), sternoclavicular joints (0-2), acromioclavicular joints (0-2), glenohumeral joints (0-2), elbows (0-2), wrists (0-2), metacarpal phalangeal joints (0-10), finger proximal interphalangeal joints (0-10), finger distal interphalangeal joints (0-8), hips (0-2), knees (0-2), ankles (0-2), tarsus/midfoot (0-2), metatarsal phalangeal joints (0-10), toe proximal interphalangeal joints (0-10).
12. Status-post complete Covid vaccination defined as at least 2 weeks after complete vaccination series.

Exclusion Criteria:

1. Pregnancy or lactation
2. Known allergic reactions to components of methotrexate or folic acid.
3. Treatment with another investigational drug or other intervention within 1 month.
4. History of chronic infection such as hepatitis and HIV. Patients with acute infection will have enrollment deferred until the infection resolves.
5. Current signs or symptoms of uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic or cerebral disease.
6. Patients with a current diagnosis of class III or IV CHF.
7. History of lymphoproliferative disease including lymphoma.
8. Overt or laboratory evidence of immunodeficiency syndromes.
9. Any opportunistic infections, including but not limited to evidence of active cytomegalovirus, active Pneumocystis carinii, aspergillosis, histoplasmosis or atypical mycobacterium infection, within the previous 6 months at screening visit.
10. History of substance abuse (drug or alcohol) within the previous 2 years.
11. Intra-articular, soft tissue or intra-muscular corticosteroid injection during the 4 weeks prior to screening.
12. History of prior use of methotrexate or biologic therapy.
13. Evidence of active infection with fever >38°
14. Current use of any other disease modifying arthritis medication including but not limited to sulfasalazine, methotrexate, hydroxychloroquine, leflunomide, or biologics in the previous 2 months. Patients on stable doses of prednisone up to 10 mg per day for at least 4 weeks prior to enrollment may participate. Non-steroidal anti-inflammatories (NSAIDS) and acetaminophen are permitted for pain during the study.
15. Hematuria or proteinuria on urinalysis.
16. The presence of anti-cyclic citrullinated peptide (Anti-CCP) antibodies >2 times the upper limit of normal.
17. For patients who participate in synovial biopsy substudy the following additional exclusion criteria apply:

1. Known prior reactions or allergies to local anesthetics or antibiotics (specifically bupivocaine, lidocaine, or cephalexin) 2. Preexisting advanced structural or functional damage to joint of interest such as prior history of trauma requiring orthopedic surgery and hardware placement, and presence of prosthetic devices (artificial joints, pacemakers, other implantable devices) 3. History of diabetes, skin infections (cellulitis), bleeding disorders, deep vein thrombosis, pulmonary embolism, history or active cancer of any kind 4. Use of blood thinners (anticoagulants) 5. History of or current chronic pain syndrome such as fibromyalgia, chronic back pain, migraines, and history of current complex regional pain syndrome, and /or current or past chronic opiate treatment 6. Significant other comorbidities and /or medication use which in physician's clinical judgment may pause procedure or post-procedure complication risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of oral methotrexate treatment versus placebo for 6 months in chronic CHIKV arthritis. | up to 6 months
  An improvement in the Disease Activity Score-28 response. The DAS-28 is a composite measure including a tender and swollen joint joint of 28 joints, patient reported disease severity measures, and the c-reactive protein

SECONDARY OUTCOMES:
Inflammation in the synovial tissue measured by synovial inflammatory cell infiltration | Up to 6 weeks
  The investigators hypothesize that treatment with methotrexate versus placebo will decrease synovial macrophage and T-cell accumulation.
Inflammatory cytokine levels in synovial tissue | Up to 6 weeks
  The investigators hypothesize that treatment with methotrexate versus placebo will dampen production of pathogenic cytokines like with TNF, IL-6, and MCP-1

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica de la Costa, Barranquilla, Colombia